CLINICAL TRIAL: NCT05706207
Title: A Phase Ia,Single Center,Open-label,Dose-escalation Study to Evaluate the Safety and Pharmacokinetics of HB0030 Injection in Patients With Advanced Solid Tumors
Brief Title: A Study of HB0030 Injection in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HB0030-01
Record Dates: First submitted 2023-01-06; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Subjects were enrolled from low to high doses. The dose groups were 0.03 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg, 10 mg/kg, 20 mg/kg, 30 mg/kg and 40 mg/kg, a total of 8 dose levels.For the first dose group (0.03mg/kg), the dose was increased according to the principle of accelerated titration combined with 3+3 dose acceleration.from 0.3mg/kg dose group,the study will adopt the 3+3 dose acceleration principle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Arm 1 (Experimental): Treatment with 0.03 mg/kg HB0030 injection administered intravenously
  Interventions: Drug: HB0030 injection
- Arm 2 (Experimental): Treatment with 0.3 mg/kg HB0030 injection administered intravenously
  Interventions: Drug: HB0030 injection
- Arm 3 (Experimental): Treatment with 1 mg/kg HB0030 injection administered intravenously
  Interventions: Drug: HB0030 injection
- Arm 4 (Experimental): Treatment with 3 mg/kg HB0030 injection administered intravenously
  Interventions: Drug: HB0030 injection
- Arm 5 (Experimental): Treatment with 10 mg/kg HB0030 injection administered intravenously
  Interventions: Drug: HB0030 injection
- Arm 6 (Experimental): Treatment with 20 mg/kg HB0030 injection administered intravenously
  Interventions: Drug: HB0030 injection
- Arm 7 (Experimental): Treatment with 30 mg/kg HB0030 injection administered intravenously
  Interventions: Drug: HB0030 injection
- Arm 8 (Experimental): Treatment with 40 mg/kg HB0030 injection administered intravenously
  Interventions: Drug: HB0030 injection

INTERVENTIONS:
Drug: HB0030 injection — 0.03 mg/kg intravenously, every 3 weeks, till tumor progress or intolerance
  Other Names: Recombinant Humanized Anti-TIGIT Monoclonal Antibody
  Arms: Arm 1
Drug: HB0030 injection — 0.3 mg/kg intravenously, every 3 weeks, till tumor progress or intolerance
  Other Names: Recombinant Humanized Anti-TIGIT Monoclonal Antibody
  Arms: Arm 2
Drug: HB0030 injection — 1 mg/kg intravenously, every 3 weeks, till tumor progress or intolerance
  Other Names: Recombinant Humanized Anti-TIGIT Monoclonal Antibody
  Arms: Arm 3
Drug: HB0030 injection — 3 mg/kg intravenously, every 3 weeks, till tumor progress or intolerance
  Other Names: Recombinant Humanized Anti-TIGIT Monoclonal Antibody
  Arms: Arm 4
Drug: HB0030 injection — 10 mg/kg intravenously, every 3 weeks, till tumor progress or intolerance
  Other Names: Recombinant Humanized Anti-TIGIT Monoclonal Antibody
  Arms: Arm 5
Drug: HB0030 injection — 20 mg/kg intravenously, every 3 weeks, till tumor progress or intolerance
  Other Names: Recombinant Humanized Anti-TIGIT Monoclonal Antibody
  Arms: Arm 6
Drug: HB0030 injection — 30 mg/kg intravenously, every 3 weeks, till tumor progress or intolerance
  Other Names: Recombinant Humanized Anti-TIGIT Monoclonal Antibody
  Arms: Arm 7
Drug: HB0030 injection — 40 mg/kg intravenously, every 3 weeks, till tumor progress or intolerance
  Other Names: Recombinant Humanized Anti-TIGIT Monoclonal Antibody
  Arms: Arm 8

SUMMARY:
This is a phase Ia single-center, open-label, dose escalation study.The objectives of this study are to evaluate the safety, toxicity, tolerability, pharmacokinetics/pharmacodynamics(PK/PD), immunogenicity, biomarkers, and antitumor activity of HB0030 in advanced solid tumor subjects.

DETAILED DESCRIPTION:
The phase Ia study will enroll up to 19-36 subjects with advanced solid tumor who have progressing tumor after standard therapy and have no better treatment option.The conventional 3+3 design will be applied for dose escalation.This study will set up 8 dose groups.HB0030 injection is administered once every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Age ≥ 18 years.
* Patients with histologically or cytologically confirmed advanced malignant solid tumor who have been intolerant of all standard therapies or recurrence after all standard therapies, and there is no better treatment option.
* At least one measurable tumor lesion According to RECIST criteria v1.1
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1
* Life expectancy ≥3 months
* Adequate organ function defined as:（No blood transfusion or hematopoietic stimulator treatment within 14 days before screening）

  1. Adequate Hematological function defined as:

     1. Absolute neutrophil count ≥1.5×109/L
     2. Platelet count≥75×109/L
     3. Hemoglobin ≥ ≥90g/L
  2. Adequate hepatic function defined as:

     1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
     2. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN; AST or ALT ≤ 5 × ULN if subjects have liver metastases or liver cancer
  3. Adequate renal function defined as:

     creatinine clearance (CrCL) > 50 mL/min (calculated by Cockcroft-Gault Equation).
  4. Adequate Coagulation function defined as:

     1. Activated partial thromboplastin time (APTT) ≤1.5×ULN
     2. International Normalized Ratio (INR)≤1.5×ULN
  5. Urine protein: qualitative urine protein ≤ 1+ or qualitative urine protein≥ 2+,24h urine protein<1g
* The fertile subjects (male and female) must agree to use reliable contraceptive methods (hormone or barrier method or abstinence) with their partners during the test period and at least 90 days after the last medication; The blood or urine pregnancy test of female patients of childbearing age within 7 days before the first administration must be negative
* Subjects can fully understand this study and voluntarily sign the informed consent form before the trial, and are willing and able to follow the clinical research and follow-up visit process.

Exclusion Criteria:

* Symptomatic central nervous system(CNS) metastases; or there is other evidence that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, which is not suitable for enrollment according to the judgment of the investigator; or patients with asymptomatic CNS metastases who are radiologically and neurologically stable > 4 weeks following CNS directed therapy, and are on a stable or decreasing dose of corticosteroids equivalent to < 10 mg prednisone/day for at least 2 weeks prior to study treatment are eligible for study entry.
* Active autoimmune disease or history of autoimmune disease requiring systemic therapy < 2 years prior to screening except hypothyroidism, vitiligo, Grave's disease, Hashimoto's disease, or Type I diabetes. Patients with childhood asthma or atopy that has not been active in the 2 years prior to study screening are eligible.
* History of Grade 3-4 immune-related adverse events (irAEs) or irAEs requiring discontinuation of prior therapies, (except for grade 3 endocrinopathy that is managed with hormone replacement therapy).
* Use of systemic corticosteroids in a dose equivalent to > 10 mg/day of prednisone or other immunosuppressive agent < 2 weeks prior to screening; the use of topical, intraocular, intra-articular, intranasal or inhaled corticosteroids (systemic absorption is low) will be allowed to prevent (e.g. allergy to contrast agents) or treat non-autoimmune condition (e.g. delayed hypersensitivity caused by exposure to allergens)
* Patients who Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

  1. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events of grade 3 or above occurred within 6 months before enrollment
  2. Serious cardiac rhythm or conduction abnormality, such as ventricular arrhythmia requiring clinical intervention, II-III degree atrioventricular block, QTcF≥450 ms, etc
  3. New York Heart Association（NYHA）cardiac function grade ≥ Grade II or left ventricular ejection fraction(LVEF)<50%
  4. Uncontrolled arterial hypertension even after standard treatment (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg)
* Uncontrolled diabetes mellitus with hemoglobin A1c > 8%.
* Patients who Have received TIGIT inhibitor treatment in the past
* Patients who Have received chemotherapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor drugs within 4 weeks before enrollment， Except for the following：

  1. Nitrosourea or mitomycin C within 6 weeks before the first use of the study drug
  2. Oral fluorouracil and small molecule targeted drugs are taken 2 weeks before the first use of the study drug or within 5 half-life of the drug(according to whichever is longer)
  3. The Chinese medicine with anti-tumor indication is within 2 weeks before the first use of the study drug
* Patients who Have received stem cell, bone marrow or solid organ transplantation in the past
* Any of the following infections：

  1. Active infection within 2 weeks before screening, requiring intravenous medication
  2. Active tuberculosis (via medical history).
  3. Positive test for HIV antibody at screening.
  4. Active hepatitis B or C. HBV carriers without active disease (HBV DNA titer < 1000 cps/mL or 200 IU/mL), or cured Hepatitis C (negative hepatitis C virus RNA test) may be enrolled.
* patients who have received major surgical treatment (excluding diagnostic puncture, venous catheterization, etc.), interventional treatment, radiotherapy and ablation treatment within 4 weeks before screening
* patients who have a history of severe allergy, has experienced 3-4 grade allergic reaction when receiving other monoclonal antibodies, or is known to be allergic to protein drugs or recombinant proteins or HB0030 drug components
* Patients who have received live virus vaccine within 30 days before screening except for Corona Virus Disease 2019(COVID-19) vaccine
* Pregnant or breast-feeding females
* Patient who has participated in other clinical studies and received study drugs within 30 days before the first dose Administration of study.
* Any other serious diseases (e.g. active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe symptoms and signs of blood coagulation disorder, heart disease).or in the judgment of the Investigator, there are some situation may interfere with the planned staging, treatment and follow-up. Or The patient's compliance is affected or the subject is at high risk of treatment complications.
* COVID-19 infected persons with positive quantitative real time(qRT) polymerase chain reaction(PCR )and/or serological test results during screening.
* Severe dyspnea or pulmonary dysfunction or need for continuous supportive oxygen inhalation.
* The skin wound, surgical site, wound site, mucosa serious ulcer or fracture did not fully heal, and the investigator judged that it was not suitable for enrollment.
* Patients with gastrointestinal bleeding within 12 weeks before the administration of the first study drug or with active gastrointestinal bleeding judged by the investigator.
* Patients with a history of interstitial lung disease or non-infectious pneumonia, except those caused by radiotherapy (enrollment shall be determined after discussion with the medical supervisor)
* Inability to comply with study and follow-up procedures
* Patients unable to comply with study procedures
* Patients who in the judgement of the Investigator are not suited to participate in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity(DLT) | Up to 21 days
  * DLT refers to the following toxicity related to HB0030 occurred during the DLT evaluation period (the first treatment cycle):
    1. Hematological Dose Limiting toxicity include：
       1. Grade 4 anaemia
       2. Grade IV neutropenia confirmed by reexamination.
       3. Grade 3 or higher febrile neutropenia
       4. Grade 4 thrombocytopenia or grade 3 thrombocytopenia with bleeding
    2. Nonhematologic Dose Limiting toxicity include：
       1. Grade IV Nonhematologic Toxicity
       2. Grade 3 non-hematological toxicity, which cannot be recovered to ≤ Grade 2 within 3 days after the best treatment
       3. Failure to control grade III hypertension (uncontrolled <160/100 mmHg in 7 days with appropriate antihypertensive therapy)
       4. Other toxicities judged by investigators to require permanent discontinuation of HB0030
  * the above toxic reaction is evaluated by laboratory ,physical ,ECG, radiographic examination and etc.
  * Adverse events will be graded by NCI CTCAE v5.0
Maximum Tolerated Dose(MTD) | Up to 24 Months
  - Maximum Tolerated Dose is defined as the highest dose in which the number of cases of DLT is less than 1/3 of the total patients in the first treatment cycle (DLT evaluation period) of the dose increasing stage.Six subjects are required to confirm MTD

SECONDARY OUTCOMES:
Maximum serum concentration(Cmax) | within 48 hours after single HB0030 administered
  * Cmax refers to The maximum blood concentration of HB0030 after administration.
  * Sample concentration analysis method adopts ELISA .
  * parameters will be calculated by Phoenix WinNonlin version 8.3 using noncompartmental analysis
half-life (t1/2) | within 3 months after first dose of HB0030 administered
  * t1/2 refers to time of a half reduction of total drug concentration in Body.
  * parameters will be calculated by Phoenix WinNonlin version 8.3 using noncompartmental analysis
time of maximum concentration(Tmax) | within 48 hours after single HB0030 administered
  - peak time after HB0030 administration.parameters will be calculated by Phoenix WinNonlin version 8.3 using noncompartmental analysis
AUClast | Up to 24 Months
  * AUClast refers to Area under the curve (AUC) from the time of 0 to the last measurable concentration.
  * parameters will be calculated by Phoenix WinNonlin version 8.3 using noncompartmental analysis.
Objective response rate (ORR) | Up to 24 Months
  ORR defined as the number of patients were confirmed complete response(CR) and/or partial response(PR) according to RECIST 1.1 divided by the patients with at least one tumour evaluation
Disease control rate (DCR) | Up to 24 Months
  DCR defined as the number of patients were confirmed CR and/or PR and/or stable disease(SD) according to RECIST 1.1 divided by the patients with at least one tumour evaluation
Duration of response (DOR) | Up to 24 Months
  DOR defined as time from the first record of CR or PR to the first record of disease progression or death of subjects
Anti-drug antibody (ADA) | Up to 24 Months
  Using the ELISA method to detect the anti-drug antibody production in peripheral blood after HB0030 administration.

CONTACTS AND LOCATIONS:
Overall Officials: huan zhou, master, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- the First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No